CLINICAL TRIAL: NCT03422783
Title: Correlation Between NoL Index Response to Standardized Stimulus Under General Anesthesia and: Post-operative Opioid Consumption and Pain, Pre-operative Phenotype and Pain Biomarkers
Brief Title: Correlation Between NOL Index After Stimulus and Post-operative Opioid, Pain, Pre-operative Phenotype
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped in march 2024 because lead investigator left Canada
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, Director of Research in the Department of Anesthesiology, Ciusss de L'Est de l'Île de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-1071
Record Dates: First submitted 2018-01-11; First posted 2018-02-06 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Pain, Postoperative; Anesthesia; Catastrophizing; Nociceptive Pain
Keywords: Monitoring; Biomarker; Thoracoscopy
MeSH Terms: conditions — Pain, Postoperative; Nociceptive Pain | interventions — Biomarkers

STUDY DESIGN:
Intervention Model Description: Prospective Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Included patients (Experimental): There is only one arm in this study. Intervention will be electrical forearm stimulus under general anesthesia and the response of NOL index following this stimulus and its correlation with postoperative parameters such as pain and opioid consumption in post anesthesia care unit.
  Interventions: Device: Standardized tetanic stimulation; Diagnostic Test: Catastrophizing score; Diagnostic Test: Nociceptive threshold; Biological: Biomarkers

INTERVENTIONS:
Device: Standardized tetanic stimulation — The "intervention" is not a drug, but it is standardized electrical stimulus applied with a muscle relaxation monitor on the forearm of the anesthetized patient. The NoL index is registered in response to this stimulus in an observational manner.
  Device: Device PMD200TM offering intraoperative NoL Index
Diagnostic Test: Catastrophizing score — Pre-operative catastrophizing score is correlated with post-operative pain and opioid consumption
Diagnostic Test: Nociceptive threshold — Nociceptive threshold for pressure, heat and electrical stimulation are associated with post-operative pain and will be assessed preoperatively to see if there is correlation between them and the NOL index response to the nociceptive stimulus (see intervention 1)
Biological: Biomarkers — Some biomarkers of inflammation and endogenous opioids are associated with post-operative pain. Blood samples will be withdrawn at D0 before surgery starts, D1 (H24) and D2 (H48) after surgery to see if they correlate with NOL changes after the stimulus described in intervention 1 above

SUMMARY:
This study evaluates the correlation between NoL index response to standardized stimulus under general anesthesia and the post-operative pain, assessed by opioid consumption and numerical pain scores after video-assisted thoracoscopy (VATS).

DETAILED DESCRIPTION:
The NoL index, a nociception monitor using a multiparametric approach, has shown an excellent sensitivity and specificity in detecting noxious stimuli under general anesthesia. This monitor is better than any other parameter in grading nociception under general anesthesia. More recently, it has recently been shown a strong correlation between NoL index response to nociceptive stimulus and the level of opioid analgesia during surgery. No study has evaluated that NoL could predict post-operative pain so far. It has not yet been proven that NoL was correlated with post-operative opioid consumption or with post-operative pain scores.

Some phenotypic factors were previously shown to correlate with post-operative pain and opioid consumption, such as psychological factors and tests, or also assessment of some pre-operative nociceptive thresholds (NT). Pain catastrophizing was proven in several studies to correlate with acute post-operative pain.

So far, no study compared each of these preoperative psychological factors or nociceptif thresholds to the NoL index response to intraoperative standardized pain stimulus in terms of correlation with post-operative opioid requirements and pain scores.

Moreover, there is no study evaluating the pro-inflammatory protein profiles that might likely be correlated to inter-individual differences in NoL response after this standardized nociceptive stimulus under general anesthesia.

This study will assess the level of correlation between NoL index response to standardized stimulus under general anesthesia and the post-operative pain, assessed by opioid consumption and numerical pain scores after video-assisted thoracoscopy (VATS). It also evaluates the correlation between NoL index response to standardized stimulus under general anesthesia and pre-operative phenotype and post-operative pain biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (Age 18 or older)
* ASA status I, II or III
* elective video assisted thoracoscopy under general anesthesia

Exclusion Criteria:

* history of coronary artery disease
* serious cardiac arrhythmia (including atrial fibrillation),
* history of substance abuse,
* chronic use of psychotropic and/or opioid drugs,
* use of drugs that act on the autonomic nervous system (including β-blockers),
* history of psychiatric diseases,
* allergy to any drug used in the study protocol,
* refusal of the patient
* unexpected difficult airway requesting excessive, possibly painful airway manipulations
* unexpected intraoperative complications requiring strong hemodynamic support (transfusions, vasopressors, inotropes)
* conversion to thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Correlation between NoL index and Hydromorphone consumption H24 | Day 1 at 24 hours
  Correlation between NoL index absolute values after electrical stimulus under general anesthesia and Total hydromorphone consumption (PACU and PCA) 24h after surgery

SECONDARY OUTCOMES:
Pain scores (NRS) in PACU from 0 to 10 | Day 0 at hour 2
  Pain scores from 0 to 10 after surgery, using numerical rating scale in post anesthesiology care unit
Correlation between NoL index and Pain scores (NRS from 0 to 10) in PACU | Day 0 at hour 2
  Correlation between NoL index absolute values after electrical stimulus under general anesthesia and Pain scores after surgery, in post anesthesiology care unit
Pain scores (NRS from 0 to 10) at H24 at rest | Day 1 at 24 hours
  Pain scores (NRS from 0 to 10) at H24 at rest
Correlation between NoL index and Pain scores (NRS) from 0 to 10 at H24 at rest | Day 1 at 24 hours
  Correlation between NoL index absolute values after electrical stimulus under general anesthesia and Pain scores (NRS) at H24 at rest
Pain scores (NRS) at H24 while coughing from 0 to 10 | Day 1 at 24 hours
  Pain scores (NRS) at H24 while coughing from 0 to 10
Correlation between NoL index and Pain scores (NRS) from 0 to 10 at H24 while coughing | Day 1 at 24 hours
  Correlation between NoL index absolute values after electrical stimulus under general anesthesia and Pain scores (NRS) at H24 while coughing
Pain scores (NRS) at H48 at rest from 0 to 10 | Day 2 at 48 hours
  Pain scores (NRS) at H48 at rest from 0 to 10
Correlation between NoL index and Pain scores (NRS) from 0 to 10 at H48 at rest | Day 2 at 48 hours
  Correlation between NoL index absolute values after electrical stimulus under general anesthesia and Pain scores (NRS) at H48 at rest
Pain scores (NRS) at H48 while coughing from 0 to 10 | Day 2 at 48 hours
  Pain scores (NRS) at H48 while coughing from 0 to 10
Correlation between NoL index and Pain scores (NRS) from 0 to 10 at H48 while coughing | Day 2 at 48 hours
  Correlation between NoL index absolute values after electrical stimulus under general anesthesia and Pain scores (NRS) at H48 while coughing
total hydromorphone consumption (mg) in PACU | Day 0 at 2 hours
  general anesthesia and total hydromorphone consumption (mg) in PACU
Correlation between NoL index and total hydromorphone consumption (mg) in PACU | Day 0 at 2 hours
  Correlation between NoL index absolute values after electrical stimulus under general anesthesia and total hydromorphone consumption (mg) in PACU
Total hydromorphone consumption (mg) at H48 | Day 2 at 48 hours
  Total hydromorphone consumption (mg) at H48
Correlation between NoL index and total hydromorphone consumption (mg) at H48 | Day 2 at 48 hours
  Correlation between NoL index absolute values after electrical stimulus under general anesthesia and total hydromorphone consumption (mg) at H48
Pain catastrophizing scale from 0 to 50 (fully validated and published questionnaire) | Pre-operative, 2 hours prior to surgery
  Pain catastrophizing scale from 0 to 50
Correlation between Pain catastrophizing scale from 0 to 50 and Total (hydromorphone consumption at day 1 24 hours) | Day 1 at 24 hours
  Correlation between Pain catastrophizing scale and Total hydromorphone
Correlation between Pain catastrophizing scale from 0 to 50 and NoL index | Day 0
  Correlation between pre-operative Pain catastrophizing scale and NoL index absolute values after electrical stimulus under general anesthesia
State-Trait anxiety Inventory from 0 to 80 (fully validated and published questionnaire) | Day 0
  State-Trait anxiety Inventory from 0 to 80
Correlation between State-Trait anxiety Inventory questionnaire from 0 to 80 and NoL index | Day 0
  Correlation between pre-operative State-Trait anxiety Inventory and NoL index absolute values after electrical stimulus under general anesthesia
Correlation between State-Trait anxiety Inventory from 0 to 80 and Total hydromorphone consumption at H24 | Day 1 24 hours
  Correlation between State-Trait anxiety Inventory and Total hydromorphone consumption at H24
mechanic pain threshold | Pre-operative, 2 hours prior to surgery
  mechanic pain threshold using electronic Von Frey
thermal pain threshold | Pre-operative, 2 hours prior to surgery
  thermal pain threshold using Qsense device
electrical pain threshold | Pre-operative, 2 hours prior to surgery
  electrical pain threshold using Pain Matcher device
Biomarkers level Pre-op | Pre-operative, H0 right after induction of general anesthesia
  Biomarkers level Pre-op
Biomarkers level H24 | Day 1 24 hours
  Biomarkers level H24
Biomarkers level H48 | Day 2 48 hours
  Biomarkers level H48
Brief Pain inventory (3M) Questionnaire (validated and published questionnaire) | 3 months
  Brief Pain inventory (3M)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montreal, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No